CLINICAL TRIAL: NCT05427214
Title: A Prospective Imaging Study of Target Definition and Simulation-free Planning Workflows on the Halcyon 4.0 System for Patients Receiving Radiation Therapy
Brief Title: Imaging Study on Halcyon 4.0 System for Patients Receiving Radiation Therapy
Acronym: Dragon
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Varian Medical Systems (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 202205118
Record Dates: First submitted 2022-06-16; First posted 2022-06-22 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-10

CONDITIONS: Brain Cancer; Head and Neck Cancer; Lung Cancer; Gastric Cancer; Ovarian Cancer; Colon Cancer
Keywords: radiation therapy; halcyon; brain radiation; thoracic radiation; abdominal radiation; pelvic radiation
MeSH Terms: conditions — Brain Neoplasms; Head and Neck Neoplasms; Lung Neoplasms; Stomach Neoplasms; Ovarian Neoplasms; Colonic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Halcyon 4.0 imaging (Experimental): Patients planning to receive radiation therapy to the head and neck/brain, thorax, abdomen, or pelvis will undergo imaging on the Halcyon 4.0 system. Patients will return for a minimum of 2 sessions over 9 weeks, with a cumulative total of 10 images being collected.
  Interventions: Device: Halcyon 4.0 system

INTERVENTIONS:
Device: Halcyon 4.0 system — During each of the 1 or more imaging sessions, no more than 6 images total will be acquired. Only 5 images total across all of the imaging sessions will be used toward the study endpoint.

SUMMARY:
This prospective imaging study is evaluating the feasibility of using the Halcyon 4.0 radiotherapy system for radiation therapy planning in patients with cancer. The Halcyon 4.0 system has been engineered to decrease the image acquisition time and the radiation exposure, but the system has not yet been clinically validated for use in radiation planning. This pilot study will evaluate images obtained on the Halcyon 4.0 system to assess if the quality is sufficient for radiation treatment plan construction.

ELIGIBILITY:
Eligibility Criteria:

* Planning to receive radiation therapy to one of the following sites:

  * Head and neck/brain (n=10)
  * Thorax (n=10)
  * Abdomen (n=10)
  * Pelvis (n=10)
* At least 18 years of age
* If the patient will be receiving IV contrast on study: Adequate renal function as defined by a serum creatinine < 1.4, or, for patients with chronic kidney disease, a stable serum creatinine < 2.0. Note: if no IV contrast will be administered on study, patient may enroll without creatinine level documented.
* If the patient is a woman of childbearing potential, a negative pregnancy test must be obtained. Contraceptive use is not an adequate documentation of no chance of pregnancy.
* Able to understand and willing to sign an IRB approved written informed consent document.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2022-08-19 (Actual); Primary Completion 2024-10-17 (Actual); Study Completion 2024-10-17 (Actual)

PRIMARY OUTCOMES:
Percentage of images that are of sufficient quality for patient primary treatment plan construction | At 9 weeks
  If the treatment target and surrounding organs at risk can be visualized and contoured for treatment planning purposes and a treatment plan created that meets the stated objectives ( or better than the stated objectives), then the kV CBCT images will be deemed feasible.

CONTACTS AND LOCATIONS:
Overall Officials: Pamela Samson, M.D., MPHS, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu